CLINICAL TRIAL: NCT03247478
Title: Computed Tomography (CT) Reconstruction for Axillary Lymph Node Structure: a Prospective Observational Study Evaluating Response in Axillary Lymph Nodes of Breast Cancer After Neoadjuvant Chemotherapy
Brief Title: Computed Tomography (CT) Reconstruction for Axillary Lymph Node Structure
Acronym: CTREP
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Director of Breast Center of Peking University Cancer Hospital, Peking University
Other Study IDs: BCP20
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Invasive Breast Cancer
Keywords: Computed tomography (CT) reconstruction; axillary lymph node status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Axillary lymph node status are determined in FNA/CNB and surgical specimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- invasive breast cancer: Patients with invasive breast cancer who underwent computed tomography (CT) reconstruction of axillary lymph node for assessment of lymph node response after NAC are eligible for this study. Axillary lymph node metastasis is confirmed by fine needle aspiration (FNA) or core needle biopsy (CNB) at initial diagnosis.

SUMMARY:
This is a prospective, single-center, non-randomized, non-controlled observational study.

DETAILED DESCRIPTION:
The negative predictive value of ultrasound for lymph node with neoadjuvant chemotherapy is low, magnetic resonance imaging (MRI) or PET/CT did not significantly improve specificity to axillary lymph node. The aim of this study is to determine performance of computed tomography (CT) reconstruction on evaluation of lymph node status after neoadjuvant chemotherapy in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer with axillary lymph node metastasis by confirmed by fine needle aspiration (FNA) or core needle biopsy (CNB).
* Underwent computed tomography (CT) reconstruction for assessment of axillary lymph node status before and after neoadjuvant chemotherapy (NAC).
* Attend the study voluntarily, sign the informed consent.

Exclusion Criteria:

* Contradiction for adjuvant chemotherapy.
* Contradiction for proceeding surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Invasive breast cancer with axillary lymph node metastasis: stage N1-2.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive-predictive value (PPV) and negative-predictive value (NPV) of Computed tomography (CT) reconstruction for axillary lymph node status after neoadjuvant chemotherapy. | within 6 weeks after obtaining the post-surgery pathological results
  Sensitivity, specificity, positive-predictive value (PPV) and negative-predictive value (NPV) of Computed tomography (CT) reconstruction for axillary lymph node status after neoadjuvant chemotherapy will be assessed.

SECONDARY OUTCOMES:
Rreceiver operating characteristic (ROC) curve analysis | within 6 weeks after obtaining the post-surgery pathological results
  The diagnostic performance of computed tomography (CT) reconstruction for the evaluation of ALN after NAC was evaluated with receiver operating characteristic (ROC) curve analysis. The diagnostic accuracy was estimated by calculating the area under the ROC curve.

CONTACTS AND LOCATIONS:
Overall Officials: Li-ze Wang, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China